CLINICAL TRIAL: NCT05941585
Title: A Clinical Study to Evaluate the Safety, Efficacy and Pharmacokinetics of Mitoxantrone Hydrochloride Liposome Injection Combined With Chemotherapy in Previously Untreated de Novo Acute Myeloid Leukemia
Brief Title: Mitoxantrone Hydrochloride Liposome Combined With Chemotherapy in Untreated de Novo Acute Myeloid Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023004; NCT05893329 (obsolete NCT alias)
Record Dates: First submitted 2023-07-01; First posted 2023-07-12 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-02

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mitoxantrone hydrochloride liposome injection combined with of cytarabine (Experimental): Patients will receive mitoxantrone hydrochloride liposome injection combined with standard-dose of cytarabine.
  Interventions: Drug: Mitoxantrone hydrochloride liposome injection30mg/m2; Drug: Cytarabine(standard-dose:d1-d7100mg/m2/day)
- mitoxantrone hydrochloride liposome with cytarabine and homoharringtonine (Experimental): Patients will receive mitoxantrone hydrochloride liposome injection combined with intermediate-dose of cytarabine and homoharringtonine.
  Interventions: Drug: HomoharringtonineD1-D7(2mg/m2/day); Drug: Cytarabine(intermediate-dose:d1-d4100mg/m2/day, d5-d7 1g/m2); Drug: Mitoxantrone hydrochloride liposome injection24mg/m2
- mitoxantrone hydrochloride liposome injection combined with cytarabine and venetoclax (Experimental): Patients will receive mitoxantrone hydrochloride liposome injection with cytarabine and venetoclax.
  Interventions: Drug: Mitoxantrone hydrochloride liposome injection30mg/m2; Drug: Venetoclax (d4 100mg/day, d5200mg/day ,d6-d12 400mg/day); Drug: Cytarabine(standard-dose:d1-d7100mg/m2/day)

INTERVENTIONS:
Drug: Mitoxantrone hydrochloride liposome injection30mg/m2 — Mitoxantrone hydrochloride liposome intravenous infusion on day 1 (30mg/m2)
  Arms: mitoxantrone hydrochloride liposome injection combined with cytarabine and venetoclax; mitoxantrone hydrochloride liposome injection combined with of cytarabine
Drug: HomoharringtonineD1-D7(2mg/m2/day) — Homoharringtonine intravenous infusion on D1-D7,2mg/m2/day in a 4-week treatment cycle.
  Arms: mitoxantrone hydrochloride liposome with cytarabine and homoharringtonine
Drug: Venetoclax (d4 100mg/day, d5200mg/day ,d6-d12 400mg/day) — Venetoclax d4-d12 (d4 100mg/day, d5200mg/day ,d6-d12 400mg/day)in a 4-week treatment cycle.
  Arms: mitoxantrone hydrochloride liposome injection combined with cytarabine and venetoclax
Drug: Cytarabine(standard-dose:d1-d7100mg/m2/day) — Cytarabine intravenous infusion on d1-d7 ,100mg/m2/day
  Arms: mitoxantrone hydrochloride liposome injection combined with cytarabine and venetoclax; mitoxantrone hydrochloride liposome injection combined with of cytarabine
Drug: Cytarabine(intermediate-dose:d1-d4100mg/m2/day, d5-d7 1g/m2) — d1-d4100mg/m2/day, d5-d7 1g/m2
  Arms: mitoxantrone hydrochloride liposome with cytarabine and homoharringtonine
Drug: Mitoxantrone hydrochloride liposome injection24mg/m2 — Mitoxantrone hydrochloride liposome intravenous infusion on day 1 (24mg/m2)
  Arms: mitoxantrone hydrochloride liposome with cytarabine and homoharringtonine

SUMMARY:
The purpose of this study is to determine the safety, efficacy and pharmacokinetics of mitoxantrone hydrochloride liposome injection combined with chemotherapy in previously untreated de novo acute myeloid leukemia.

DETAILED DESCRIPTION:
This is a prospective, multi-center, randomized, open-label, three-arm clinical study to explore the efficacy among three chemotherapy regimens combined with mitoxantrone hydrochloride liposome in previously untreated de novo acute myeloid leukemia. Patients will be randomized to different treatment group and be given different induction therapy in the first cycle. If patients do not achieve Morphologic Leukemia-free State (MLFS) after the first induction cycle, they will receive the second induction therapy with mitoxantrone hydrochloride liposome, cytarabine and venetoclax. Mitoxantrone hydrochloride liposome will be given on day 1 at the dose of 24 mg/m2 or 30 mg/m2 and be combined with cytarabine, venetoclax or homoharringtonine. A maximum of 2 cycles of induction therapy are planned.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the study and voluntarily sign informed consent.
2. Age: 18~65 (including 18) years old, gender unlimited.
3. Patients diagnosed with acute myeloid leukemia according to "The 2016 revision to the World Health Organization classification of myeloid neoplasms and acute leukemia" who haven't been treated.
4. Eastern Cooperative Oncology Group (ECOG) physical state score: 0-1.
5. Fit for intensive chemotherapy.
6. The function of main organs should meet the following standards before treatment:

   Kidney: Serum creatinine ≤ 1.5 × Upper limit of normal range (ULN) Liver: Total bilirubin ≤ 1.5 × ULN, AST and ALT ≤ 3× ULN
7. Patients should agree to use contraception (such as intrauterine device [IUD], contraceptive pill or condom) during the study period and within 6 months after the end of the study; Female patients must have a negative serum pregnancy test within 7 days before enrollment.

Exclusion Criteria:

1. Any of the following cases:(1) diagnosed as acute promyelocytic leukemia (APL);(2) chronic myelogenous leukemia in blast crisis;(3) AML with central nervous system leukemia.
2. AML arising from prior cytotoxic chemotherapy or radiotherapy for other tumours.
3. Patient has been previously diagnosed with another malignancy in last 5 years (except for cured basal cell carcinoma of skin or cervical carcinoma in situ).
4. Has been previously treated with doxorubicin or other anthracyclines and drugs for AML.
5. Allergic history of mitoxantrone hydrochloride injection or any other drugs used in this study.
6. Those on systemic anti-infective therapy with poorly controlled infection (signs of infection progression within 1 week prior to the first dose, or as determined by the investigator).
7. Patient who is suffering from severe hemorrhagic diseases, such as haemophilia A, haemophilia B, von Willebrand disease and any other spontaneous bleeding require medical treatment.
8. The estimated survival time is less than 3 months.
9. Any of the following conditions occurs in cardiac function:(1) Long QTc syndrome or QTc interval > 480 ms;(2) Complete left bundle branch block or severe atrioventricular block disease (without a pacemaker);(3) Serious and uncontrolled arrhythmias and unstable angina pectoris requiring drug treatment;(4) History of chronic congestive heart failure, New York Heart Association (NYHA)≥grade 3;(5) The cardiac ejection fraction is less than 50% in Echocardiography;(6)Uncontrollable hypertension (defined as multiple measurements of systolic blood pressure > 150 mmHg or diastolic blood pressure > 90 mmHg under drug control);(7) History of myocardial infarction, unstable angina pectoris, viral myocarditis or severe pericardial disease, ECG evidence of acute ischemia or active conduction system abnormalities within 6 months before first dose.
10. Patients have thromboembolic events within 6 months prior to first dose, such as cerebrovascular accidents (including transient ischemic attack) and pulmonary embolism.
11. HBsAg/HBcAb positive with HBV-DNA higher than the lower limit of the detection value of the research center , hepatitis C antibody-positive with HCV-RNA higher than the lower limit of the detection value of the research center, or HIV antibody positive in the preliminary screening.
12. Patients who have been treated with strong/moderate CYP3A inducers/inhibitors or P-gp inhibitors within 7 days prior to first dose (for treatment group 3 only).
13. Patients who cannot take oral medications or have absorption disorder (for treatment group 3 only).
14. Patient is suffering from any serious and /or non-controllable disease, or the investigator determines that the disease might affect the participation of patients in the study, including (but not limited to, uncontrolled diabetes, dialysis related kidney diseases, severe liver diseases, life-threatening autoimmune diseases and hemorrhagic diseases, drug abuse, neurological diseases, etc.).
15. Pregnant or lactating female.
16. Patients who are not suitable for this study as decided by the investigator due to other reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Up to approximately one month
  The frequency and severity of adverse events during treatment, abnormalities in vital signs, physical examinations, laboratory tests, etc

SECONDARY OUTCOMES:
Complete remission rate（CR） | Up to approximately nine weeks
  Proportion of patients with complete remission
Complete remission or complete remission with partial hematologic recovery (CR/CRh) | Up to approximately nine weeks
  Proportion of patients with complete remission or complete remission with partial hematologic recovery.
Composite remission rate (CRc) | Up to approximately nine weeks
  Proportion of subjects with complete remission (CR) or complete remission with partial hematologic recovery (CRh) or complete remission with incomplete hematologic recovery (Cri).
Minimal Residual Disease (MRD)-negative composite remission rates | Up to approximately nine weeks
  Among those who have achieved composite remission, proportion of patients who is MRD-negative.
Event-free survival (EFS) | Up to approximately 3 years.
  It is defined as the time from the start of randomization to the occurrence of induction failure or disease progression or death from any cause (whichever occurs first).
Relapse-free Survival (RFS) | Up to approximately 3 years.
  It is defined as the time from the start of achieving remission to disease progression, death from any cause or the last follow-up
Overall survival (OS) | Up to approximately 3 years.
  It is defined as the time from the start of randomization to the death from any cause.
Blood concentrations of total and free mitoxantrone. | 30 minutes before administration and 5min, 6, 24, 72, 144, 288, 432, 648 hours after administration of Mitoxantrone hydrochloride liposome on day 1
  Blood was taken to measure the required concentration at different time points

CONTACTS AND LOCATIONS:
Overall Officials: wang jianxiang, MD, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, China